CLINICAL TRIAL: NCT06311253
Title: Non-surgical Periodontal Treatment With Adjunctive Use of Lactoferrin Contained in Toothpaste and Mouthwash: Randomized Clinical Trial
Brief Title: Non-surgical Periodontal Treatment With Adjunctive Use of Lactoferrin Contained in Toothpaste and Mouthwash
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-LACTOFERRINPREGNANT
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Periodontal Diseases
Keywords: pregnant patients
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental)
  Interventions: Other: Emoform Glic Toothpaste; Other: Emoform Glic Mouthwash
- Control group (Active Comparator)
  Interventions: Other: Emoform Glic Toothpaste

INTERVENTIONS:
Other: Emoform Glic Toothpaste — Daily use of Emoform Glic toothpaste twice a day during home oral hygiene
Other: Emoform Glic Mouthwash — Daily use of Emoform Glic mouthwash twice a day during home oral hygiene
  Arms: Trial group

SUMMARY:
The aim of the study is to assess the effect of lactoferrin in LBC complex can be effective in reducing periodontal clinical parameters in a 6-month study on pregnant patients.

DETAILED DESCRIPTION:
The aim of the study is to assess the effect of lactoferrin in LBC complex can be effective in reducing periodontal clinical parameters in a 6-month study on pregnant patients. Patients' enrollment will be conducted according to inclusion criteria.

At the first visit, periodontal parameters will be recorded: Plaque Index (PI), recession (R) Bleeding on Probing (BoP), modified Marginal Gingival Index (mMGI), Papillary Marginal Gingival (PMGI), Plaque Control Record ( PCR %), Approximal Plaque Index (API), Clinical Attachment loss (CAL) and Probing Pocket Depth (PPD).

Professional debridement will be conducted with piezoelectric instrumentation and air-flow administration with glycine powders.

Subsequently, patients will be randomly divided into two groups:

- the Trial group, in which patients will perform home oral hygiene with Emoform Glic toothpaste + mouthwash twice a day the Control group, in which patients will perform home oral hygiene with Emoform Glic toothpaste twice a day.

Professional debridement will be repeated every 3 months. Periodontal indexes evaluation will be conducted at the baseline (T0), after 1 month (T1), after 3 months (T2), and after 6 months (T3).

ELIGIBILITY:
Inclusion Criteria:

* women at the 4th month of pregnancy

Exclusion Criteria:

* presence of cardiac pacemaker
* neurological and psychiatric diseases
* patients taking bisphosphonates during the previous 12 months from the - beginning of the study
* patients undergoing anticancer therapy.
* patients with poor compliance.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Recession (R) | Baseline, 1, 3 and 6 months
  Distance (in mm) between the gingival margin and the amelo-cemental junction.
Change in Plaque Index (Silness and Loe, 1964) | Baseline, 1, 3 and 6 months
  Scoring criteria:
  0 = no plaque;
  1. = thin plaque layer at the gingival margin, only detectable by scraping with a probe;
  2. = moderate layer of plaque along the gingival margin; interdental spaces free, but plaque is visible to the naked eye;
  3. = abundant plaque along the gingival margin; interdental spaces filled with plaque.
Change in Bleeding on Probing (BoP) | Baseline, 1, 3 and 6 months
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 6 sites.
  Percentage of sites with bleeding on probing determines the BOP%.
Change in Probing Pocket Depth (PPD) | Baseline, 1, 3 and 6 months
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in modified Marginal Gingival Index (mMGI) | Baseline, 1, 3 and 6 months
  Scoring criteria:
  0 = Absence of inflammation
  1. = Mild inflammation (marginal or papillary unit)
  2. = Mild inflammation (entire marginal and papillary unit)
  3. = Moderate inflammation
  4. = Severe inflammation
Change in Papillary Marginal Gingival Index (PMGI) | Baseline, 1, 3 and 6 months
  Numerical score from 0 to 3 of gingival inflammation. Papille and gingival margins (vestibular and lingual) are given a score from 0 to 3. The score is given by the total amount of inflamed sites on the total of examined sites.
Change in Plaque Control Record (PCR%) | Baseline, 1, 3 and 6 months
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.
Change in Clinical Attachment Loss (CAL) | Baseline, 1, 3 and 6 months
  Measurement (in mm) of the position of the gingival margin in relation to the cemento-enamel junction (CEJ).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data are available upon motivated request to the Principal Investigator.